CLINICAL TRIAL: NCT03092219
Title: A Randomized, Blinded, No-Treatment Control, Multicenter, Prospective Clinical Study of TEOSYAL RHA® Redensity for the Treatment of Moderate to Severe Dynamic Perioral Rhytids
Brief Title: RHA Redensity - Perioral Rhytids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teoxane SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TEO-RHA-1501
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Results first posted 2020-07-08 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Perioral Rhytids; Aging; Wrinkle
Keywords: Perioral rhytids; Dermal filler; Hyaluronic acid; Aging; Wrinkle

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- TEOSYAL RHA Redensity (Experimental): Injection of TEOSYAL RHA Redensity into the perioral lines (n=150). Up to 6.0 mL (max 3 mL for upper and max 3 mL for lower) injected into the dermis, including the superficial dermis. Touch-up treatment provided at 2 weeks.
  Interventions: Device: TEOSYAL RHA Redensity
- No Treatment (No Intervention): No treatment control group (n=52).

INTERVENTIONS:
Device: TEOSYAL RHA Redensity — A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of streptococcus zooepidemicus, formulated to a concentration of 15 mg/g and 0.3% w/w lidocaine in a physiologic buffer.
  Arms: TEOSYAL RHA Redensity

SUMMARY:
Randomized, blinded, No-Treatment control, multi-center, prospective clinical study, to identify whether TEOSYAL RHA® Redensity is more effective than No-Treatment in the correction of moderate to severe dynamic perioral rhytids at Week 8 after last treatment (i.e., initial or touch-up treatment).

The Treating Investigator (TI) at screening will evaluate the subject's perioral rhytids severity using the Perioral Rhytids Severity Rating Scale (PR-SRS) for eligibility of the subject for the study.

The Blinded Live Evaluator (BLE) at screening will evaluate the subject's perioral rhytids severity using the PR-SRS in order to confirm eligibility and to establish a pre-treatment (Baseline) score for assessment of effectiveness.

This is done independently of the TI, and exact concordance between the BLE and the TI is not necessary for eligibility of the subject in this study.

Enrolled subjects will be randomized to either the TEOSYAL RHA® Redensity treatment group or the "No-Treatment" control group (ratio 3:1).

The TI will administrate the study device, and if necessary, subjects will receive a touch-up treatment 14 days following the initial treatment to optimize the results.

The TI will conduct safety and effectiveness evaluations at study visits, which occurred at Week 4, 8, 12, 16, 24, 36, and 52 after the last treatment, (i.e., initial or touch-up treatment) and 4 weeks after a Repeat-Treatment.

The Blinded Live Evaluator (BLE) will conduct assessments of effectiveness during the trial, including assessment of the primary endpoint at Week 8 after the last treatment (i.e., initial or touch-up treatment). The BLE will conduct effectiveness evaluations at Week 8, 12, 16, 24, 36, and 52 after the last treatment (i.e., initial or touch-up treatment).

All subjects will be followed for 52 weeks after the last treatment (i.e., initial treatment or touch-up), at which point they will be offered Repeat-Treatment (provided that the TI deems the treatment to be appropriate and the subject agrees) and will be then followed for 4 weeks after Repeat-Treatment before exiting the study.

If a subject returns to his pre-treatment PR-SRS score at Week 12 or Week 16 or Week 24 or Week 36 after initial treatment or touch up (as assessed by the TI), subjects are eligible for optional Early-Retreatment if necessary at 12 or 16 or 24 or 36 weeks after last treatment (provided that the TI deems the treatment appropriate, and the subject agrees).

Subjects will be then followed for an additional 4 weeks after Repeat-Treatment.

Subjects who will receive optional Early-Retreatment at Week 12 or Week 16 or Week 24 or Week 36 after the after initial treatment or touch-up, will be offered Repeat-Treatment at Week 52.

Subjects randomized to the "No-Treatment" control group will receive their first treatment after the primary endpoint evaluation (Week 8 after randomization) and then will be followed the same schedule as the initial treatment group.

ELIGIBILITY:
Inclusion Criteria :

* Outpatient, male or female of any race, 22 years of age or older
* Moderate to severe perioral rhytids of grade 2 or 3 on the four-point PR-SRS (ranging from 0-3)
* Willing to abstain from facial aesthetic procedures/therapies that could interfere with study evaluations
* Able to follow study instructions and complete all required visits.
* Sign the IRB-approved ICF, Photographic Release Form and the Authorization for Use and release of Health and Research Study Information (HIPAA) form prior to any study- related procedures being performed.

Exclusion Criteria :

* Female subjects that are pregnant, breast-feeding or of childbearing potential and not practicing reliable birth control
* Known hypersensitivity/allergy to any component of the study devices
* Known susceptibility to keloid formation, hypertrophic scarring or clinically significant skin pigmentation disorders
* Clinically significant active skin disease within 6 months
* History of connective tissue disease

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2017-12-17 (Actual); Study Completion 2019-01-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (6):
  - Beverly Hills, California
  - Santa Monica, California
  - Coral Gables, Florida
  - Omaha, Nebraska
  - High Point, North Carolina
  - Fairfax, Virginia
- Canada (2):
  - Montreal
  - Victoria

REFERENCES:
- [Derived] Sundaram H, Shamban A, Schlessinger J, Kaufman-Janette J, Joseph JH, Lupin M, Draelos Z, Carey W, Smith S, Eaton L. Efficacy and Safety of a New Resilient Hyaluronic Acid Filler in the Correction of Moderate-to-Severe Dynamic Perioral Rhytides: A 52-Week Prospective, Multicenter, Controlled, Randomized, Evaluator-Blinded Study. Dermatol Surg. 2022 Jan 1;48(1):87-93. doi: 10.1097/DSS.0000000000003238. PMID 34608092

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 202 subjects were randomized with 150 subjects allocated to TEOSYAL RHA® Redensity and 52 subjects allocated to No-Treatment control.
Groups:
- TEOSYAL RHA Redensity: Injection of TEOSYAL RHA Redensity into the perioral lines. Up to 6.0 mL (max 3 mL for upper and max 3 mL for lower) injected into the dermis, including the superficial dermis. Touch-up treatment provided at 2 weeks (up to 6.0 mL).
  TEOSYAL RHA Redensity: A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of streptococcus zooepidemicus, formulated to a concentration of 15 mg/g and 0.3% w/w lidocaine in a physiologic buffer. It is supplied in individual treatment syringes with 30G ½ inch disposable sterile needles.
- No Treatment: No treatment control group.
Period: Overall Study
Arm/Group | TEOSYAL RHA Redensity | No Treatment
Started (Randomized) | 150 | 52
Baseline / ITT Population (Visit 1 - Week 0) | 150 | 51 (Subject randomized to No Treatment group but received treatment at Visit 1.)
Primary Analysis Endpoint (Visit 4 - Week 8 after last treatment) | 150 | 51
Pooled SAFT Population (Visit 8 - Week 36 after last treatment) | 150 | 50 (2 subjects did not receive treatment at Visit 1b.)
Completed (Per Protocol Population) | 143 | 48
Not Completed | 7 | 4
Not completed — Protocol Violation | 7 | 4

BASELINE CHARACTERISTICS:
Population: One subject randomized to No-Treatment control group (n initial =52) received, due to site error, injections with TEOSYAL RHA Redensity. This subject was only included in the SAFT population and censored of the effectiveness analysis. This resulted in an ITT population of 201 subjects (TEOSYAL RHA Redensity n=150, and no Treatment control n=51).
Groups:
- Total: Total of all reporting groups
Arm/Group | TEOSYAL RHA Redensity | No Treatment | Total
Number analyzed (Participants) | 150 | 51 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (7.2) | 60.7 (7.6) | 61.4 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 50 | 197
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 10 | 35
  Not Hispanic or Latino | 125 | 41 | 166
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 143 | 51 | 194
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 29 | 9 | 39
  United States | 121 | 42 | 163
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick scale is a numerical classification schema for human skin color.
  Type I - always burns, never tans (pale white; blond or red hair; blue eyes; freckles).
  Type II - usually burns, tans minimally (white; fair; blond or red hair; blue, green, or hazel eyes) Type III - sometimes mild burn, tans uniformly (cream white; fair with any hair or eye color) Type IV - burns minimally, always tans well (moderate brown) Type V - very rarely burns, tans very easily (dark brown) Type VI - Never burns, never tans (deeply pigmented dark brown to darkest brown)
  Participants
    Type I - III | 110 | 36 | 146
    Type IV - VI | 40 | 15 | 55
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.3 (4.6) | 24.8 (4.9) | 25.1 (4.7)
Smoking History [Count of Participants; unit: Participants] — Population: This demographic variable only count the population with a smoking history. 143 from 150 participants have a smoking history in the RHA Redensity (7 missing values).
  50 from 51 participants have a smoking history in the no-treatment group (1 missing value).
  Participants
    Smoke past 5 yrs - No: number analyzed (Participants) | 143 | 50 | 193
    Smoke past 5 yrs - No | 120 | 41 | 161
    Smoke past 5 yrs - Yes: number analyzed (Participants) | 143 | 50 | 193
    Smoke past 5 yrs - Yes | 23 | 9 | 32
    Smoke currently - No: number analyzed (Participants) | 143 | 50 | 193
    Smoke currently - No | 123 | 45 | 168
    Smoke currently - Yes, ≤1 pack equivalents/day: number analyzed (Participants) | 143 | 50 | 193
    Smoke currently - Yes, ≤1 pack equivalents/day | 20 | 4 | 24
    Smoke currently - Yes, ≥1 pack equivalents/day: number analyzed (Participants) | 143 | 50 | 193
    Smoke currently - Yes, ≥1 pack equivalents/day | 0 | 1 | 1
Sun Exposure [Count of Participants; unit: Participants] — Population: 143 from 150 participants have a Sun exposure in the RHA Redensity (7 missing values).
  50 from 51 participants have a Sun exposure in the no-treatment group (1 missing values).
  Participants
    Protects face : Never: number analyzed (Participants) | 143 | 50 | 193
    Protects face : Never | 6 | 2 | 8
    Protects face : Sometimes: number analyzed (Participants) | 143 | 50 | 193
    Protects face : Sometimes | 31 | 12 | 43
    Protects face : Usually: number analyzed (Participants) | 143 | 50 | 193
    Protects face : Usually | 42 | 10 | 52
    Protects face : Always: number analyzed (Participants) | 143 | 50 | 193
    Protects face : Always | 64 | 26 | 90
    Artificial Tanning : None: number analyzed (Participants) | 143 | 50 | 193
    Artificial Tanning : None | 131 | 43 | 174
    Artificial Tanning : ≤1per session/month: number analyzed (Participants) | 143 | 50 | 193
    Artificial Tanning : ≤1per session/month | 11 | 4 | 15
    Artificial Tanning : ≥1 per session/month: number analyzed (Participants) | 143 | 50 | 193
    Artificial Tanning : ≥1 per session/month | 0 | 3 | 3
Alcohol History [Count of Participants; unit: Participants] — Population: 143 from 150 participants have an alcohol history in the RHA Redensity (7 missing values).
  50 from 51 participants have an alcohol history in the no-treatment group (1 missing values).
  Participants
    Alcohol past 5 yrs : No: number analyzed (Participants) | 143 | 50 | 193
    Alcohol past 5 yrs : No | 36 | 7 | 43
    Alcohol past 5 yrs : Yes: number analyzed (Participants) | 143 | 50 | 193
    Alcohol past 5 yrs : Yes | 107 | 43 | 150
    Alcohol currently : No: number analyzed (Participants) | 143 | 50 | 193
    Alcohol currently : No | 38 | 8 | 46
    Alcohol currently : Yes, ≤1 drink per day: number analyzed (Participants) | 143 | 50 | 193
    Alcohol currently : Yes, ≤1 drink per day | 101 | 40 | 141
    Alcohol currently : Yes, ≥ 1 drink per day: number analyzed (Participants) | 143 | 50 | 193
    Alcohol currently : Yes, ≥ 1 drink per day | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Perioral Rhytids Severity Rating Scale (PR-SRS) Score Rated by the Blinded Live Evaluator (BLE) at Week 8 After Last Treatment.
Description: The PR-SRS is a validated 4-point static scale for assessing perioral rhytids severity. Possible scores range from 0 (Absent) to 3 (Severe).
  Change = (Week 8 - Baseline score).
  A PR-SRS change of 1-grade will be considered clinically significant. The No-Treatment control group after treatment was not pooled for this primary outcome measure.
Time Frame: Week 8 after last treatment
Population: The Intent-to-Treat Population was used for this analysis. The ITT Population consisted of all subjects randomized in the TEOSYAL RHA® Redensity group and all subjects randomized in the No-Treatment control group (with the notable exception of 1 subject who received treatment with study device at Visit 1 and was censored from the ITT).
Measure: Count of Participants; unit: Participants
Arm/Group | TEOSYAL RHA Redensity | No Treatment
Number analyzed (Participants) | 150 | 51
Participants
  Responder | 121 | 4
  Not Responder | 29 | 47
Statistical Analysis 1: Comparison: TEOSYAL RHA Redensity vs No Treatment; Test type: Superiority; p = 0.0001, Fisher Exact; For this outcome measure, missing data were imputed using a LOCF (Last Observation Carried Forward) method

2. Secondary Outcome: Subject's Perception of Treatment Effectiveness as Per the FACE-Q Scale (Perioral Rhytid Domain) Questionnaire at Baseline, Weeks 4 and 8 After Last Treatment.
Description: The FACE-Q measures the experience and outcomes of aesthetic facial procedures from the patient's perspective.
  The FACE-Q questionnaire is composed of 6 questions with a score linked to answers (1 being 'Not at all' and 4 being 'Extremely').
  To calculate the FACE-Q score, outcomes from all 6 questions were pooled, data were transformed so that higher scores reflected a superior outcome and adapted to a 100- unit scale.
  The No-Treatment control group after treatment was not pooled for this secondary outcome measure.
Time Frame: Baseline, Weeks 4 and 8 after last treatment
Population: The Intent-to-Treat Population (n=150 for the TEOSYAL RHA Redensity group and n=51 for the No treatment group) was used for this analysis. Numbers of patients analyzed correspond to patients that have completed the visits and for which data were available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TEOSYAL RHA Redensity | No Treatment
Number analyzed (Participants) | 150 | 51
score on a scale
  Baseline Face-Q Score: number analyzed (Participants) | 149 | 51
  Baseline Face-Q Score | 23.3 (20.8) | 24.2 (20.2)
  Week 4 Face-Q Score: number analyzed (Participants) | 146 | 48
  Week 4 Face-Q Score | 70.0 (23.8) | 24.0 (21.5)
  Face-Q Change from Baseline to Week 4: number analyzed (Participants) | 145 | 48
  Face-Q Change from Baseline to Week 4 | 46.5 (27.3) | 0.3 (11.5)
  Week 8 Face-Q Score: number analyzed (Participants) | 147 | 49
  Week 8 Face-Q Score | 68.9 (24.3) | 21.1 (20.1)
  Face-Q Change from Baseline to Week 8: number analyzed (Participants) | 146 | 49
  Face-Q Change from Baseline to Week 8 | 45.6 (26.4) | -3.8 (12.1)

3. Secondary Outcome: Number of Subjects Who Scored Themselves Either "Much Improved" or "Improved" on Global Aesthetic Improvement (GAI) Scale at Week 8 and 4 After Last Treatment.
Description: The Global Aesthetic Improvement (GAI) is a subjective, balanced, 5-point dynamic scale assessing cosmetic improvement.
  Possible scores range from "much improved", "improved", "no change", "worse", to "much worse".
  The GAI will be assessed using the pre-injection baseline photograph. The No-Treatment control group after treatment was not pooled for this secondary outcome measure.
Time Frame: Weeks 4 and 8 after last treatment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | TEOSYAL RHA Redensity | No Treatment
Number analyzed (Participants) | 150 | 51
Participants
  Week 4: Improved | 144 | 1
  Week 4: No Improvement | 2 | 46
  Week 4: Missing values | 4 | 4
  Week 8: Improved | 141 | 0
  Week 8: No Improvement | 6 | 49
  Week 8: Missing values | 3 | 2

4. Secondary Outcome: Number of Subjects Scored Either "Much Improved" or "Improved" on Global Aesthetic Improvement (GAI) Scale by the Blinded Live Evaluator (BLE) at Week 8 After Last Treatment.
Description: as for outcome 3
Time Frame: Week 8 after last treatment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | TEOSYAL RHA Redensity | No Treatment
Number analyzed (Participants) | 150 | 51
Participants
  Improved | 135 | 4
  No Improvement | 11 | 44
  Missing values | 4 | 3

5. Secondary Outcome: Number of Subjects "Satisfied" or "Very Satisfied" With Study Treatment Using the Subject Satisfaction Scale at Week 8 After Last Treatment.
Description: The Subject Satisfaction Scale is a subjective, balanced, 5-point scale assessing subject satisfaction with study treatment. Possible scores range from with 1 (very satisfied) to 5 (very dissatisfied).
  The No-Treatment control group after treatment was not pooled for this secondary outcome measure.
Time Frame: Week 8 after last treatment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | TEOSYAL RHA Redensity | No Treatment
Number analyzed (Participants) | 150 | 51
Participants
  Satisfied | 133 | 4
  Not Satisfied | 14 | 39
  Missing values | 3 | 8

6. Secondary Outcome: Number of Participants With Adverse Events for the Safety Evaluation of TEOSYAL RHA® Redensity.
Description: The Treating Investigator will assess adverse events and record details of seriousness, severity, duration, and action taken with the study device, and relationship to the study device. AEs will be reported from the time of consent until week 52 or to 1 month following the last treatment.
Time Frame: Baseline through Week 52 following the last treatment and 4 weeks following re-treatment
Measure: Count of Participants; unit: Participants
Groups:
- SAFT Population: The SAFT Population consisted of all subjects who were randomized and received at least one treatment with the study device during the course of the study (i.e. all subjects in the No-Treatment control group and all subjects in the TEOSYAL RHA® Redensity treatment group).
  Of the 202 randomized subjects, 2 subjects did not receive any treatment during the whole study, resulting in a SAFT population of n=200.
  It is to be remembered that subjects randomized to the "No-Treatment" control group received their first treatment after the primary endpoint evaluation (Week 8 after randomization) and then followed the same schedule as the initial TEOSYAL RHA® Redensity treatment group.
Arm/Group | SAFT Population
Number analyzed (Participants) | 200
Participants
  Any Treatment Emergent Adverse Event | 120
  Any Treatment Related Adverse Event | 73
  Any Serious Adverse Event | 7
  Any Treatment Related Serious Adverse Event | 0
  Any Unexpected Adverse Device Effects | 0

7. Secondary Outcome: Number of Post-Injection Treatment Responses (From Common Treatment Responses (CTR) Diary) for the Safety Evaluation of TEOSYAL RHA® Redensity.
Description: The subjects will receive a diary booklet and instructions for recording his/her observations of the Common Treatment Responses of the study treatments for the first 14 days after treatment. The diary will be discussed during telephone follow-up visit. Subjects should complete the diary at approximately the same time each day (i.e., am or pm).
  The subject diary captures the following Common Treatment Responses (CTR) that occur following the injection of a dermal filler; specifically, redness, pain, tenderness, firmness, swelling, lumps/bumps, bruising, itching, discoloration, and "other".
  The 14-day patient CTR diary includes a detailed glossary describing all signs/symptoms listed in the diary; an option was provided to rate "other" if the subject experienced a sign/symptom that is not listed.
  The table presents the number of subjects experiencing at least 1 Common Treatment Response (CTR).
Time Frame: During 14 days after initial treatment and touch-up (2 weeks)
Population: All numbers are based on the number of total number of subjects who provided diary answers after their treatment.
Measure: Number; unit: number of subjects
Arm/Group | SAFT Population
Number analyzed (Participants) | 200
number of subjects
  Initial Treatment : Redness: number analyzed (Participants) | 199
  Initial Treatment : Redness | 131
  Initial Treatment : Pain: number analyzed (Participants) | 199
  Initial Treatment : Pain | 54
  Initial Treatment : Tenderness: number analyzed (Participants) | 199
  Initial Treatment : Tenderness | 105
  Initial Treatment : Firmess: number analyzed (Participants) | 199
  Initial Treatment : Firmess | 115
  Initial Treatment : Swelling: number analyzed (Participants) | 199
  Initial Treatment : Swelling | 146
  Initial Treatment : Lumps/Bumps: number analyzed (Participants) | 199
  Initial Treatment : Lumps/Bumps | 115
  Initial Treatment : Bruising: number analyzed (Participants) | 199
  Initial Treatment : Bruising | 154
  Initial Treatment : Itching: number analyzed (Participants) | 199
  Initial Treatment : Itching | 31
  Initial Treatment : Discoloration: number analyzed (Participants) | 199
  Initial Treatment : Discoloration | 94
  Touch-up Treatment : Redness: number analyzed (Participants) | 137
  Touch-up Treatment : Redness | 85
  Touch-up Treatment : Pain: number analyzed (Participants) | 137
  Touch-up Treatment : Pain | 29
  Touch-up Treatment : Tenderness: number analyzed (Participants) | 137
  Touch-up Treatment : Tenderness | 54
  Touch-up Treatment : Firmess: number analyzed (Participants) | 137
  Touch-up Treatment : Firmess | 57
  Touch-up Treatment : Swelling: number analyzed (Participants) | 137
  Touch-up Treatment : Swelling | 84
  Touch-up Treatment : Lumps/Bumps: number analyzed (Participants) | 137
  Touch-up Treatment : Lumps/Bumps | 59
  Touch-up Treatment : Bruising: number analyzed (Participants) | 137
  Touch-up Treatment : Bruising | 82
  Touch-up Treatment : Itching: number analyzed (Participants) | 137
  Touch-up Treatment : Itching | 11
  Touch-up Treatment : Discoloration: number analyzed (Participants) | 137
  Touch-up Treatment : Discoloration | 39

8. Secondary Outcome: Assessment of Injection Site Pain Felt by the Patient for the Safety Evaluation of TEOSYAL RHA® Redensity.
Description: The Injection Site Pain (during injection and post-injection) will be self-assessed by the subject using a 100 mm Visual Analog Scale (VAS).
  VAS is a 100 mm Visual Analog Scale with 0 meaning no pain and 100 meaning intolerable pain.
Time Frame: Baseline, Weeks 2, 12, 16, 24, 36 and 52
Population: All numbers are based on the total number of subjects where the data were available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAFT Population
Number analyzed (Participants) | 200
score on a scale
  Baseline VAS pain score during injection | 19.9 (19.7)
  Baseline VAS pain score 15 minutes after | 3.1 (8.3)
  Week 2 VAS pain score during injection: number analyzed (Participants) | 137
  Week 2 VAS pain score during injection | 25.4 (23.3)
  Week 2 VAS pain score 15 minutes after: number analyzed (Participants) | 137
  Week 2 VAS pain score 15 minutes after | 4.4 (10.1)
  Week 12 VAS pain score during injection: number analyzed (Participants) | 6
  Week 12 VAS pain score during injection | 14.3 (10.8)
  Week 12 VAS pain score 15 minutes after: number analyzed (Participants) | 6
  Week 12 VAS pain score 15 minutes after | 2.0 (4.9)
  Week 16 VAS pain score during injection: number analyzed (Participants) | 4
  Week 16 VAS pain score during injection | 25.0 (20.2)
  Week 16 VAS pain score 15 minutes after: number analyzed (Participants) | 4
  Week 16 VAS pain score 15 minutes after | 0.8 (1.5)
  Week 24 VAS pain score during injection: number analyzed (Participants) | 9
  Week 24 VAS pain score during injection | 24.8 (28.3)
  Week 24 VAS pain score 15 minutes after: number analyzed (Participants) | 9
  Week 24 VAS pain score 15 minutes after | 2.7 (6.3)
  Week 36 VAS pain score during injection: number analyzed (Participants) | 16
  Week 36 VAS pain score during injection | 40.6 (23.6)
  Week 36 VAS pain score 15 minutes after: number analyzed (Participants) | 16
  Week 36 VAS pain score 15 minutes after | 5.6 (6.2)
  Week 52 VAS pain score during injection: number analyzed (Participants) | 143
  Week 52 VAS pain score during injection | 19.7 (21.9)
  Week 52 VAS pain score 15 minutes after: number analyzed (Participants) | 143
  Week 52 VAS pain score 15 minutes after | 3.6 (10.8)

9. Secondary Outcome: Assessments of the Lip Function (Lip Movement) by the Treating Investigator (TI) for the Safety Evaluation of TEOSYAL RHA® Redensity.
Description: This Lip functionality testing was conducted by the Treating Investigator (TI) at each follow-up visit and pre- and post-injection at each injection, which occurred at Baseline, Weeks 2, 4, 8, 12, 16, 24, 36, and 52 after the last treatment.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 36, and 52 after the last treatment, (i.e., initial or touch-up treatment) and 4 weeks after a Repeat-Treatment.
Population: All percentages are based on the total number of subjects where the data were available.
Measure: Mean (Standard Deviation); unit: Proportion of words pronounced correctly
Arm/Group | SAFT Population
Number analyzed (Participants) | 200
Proportion of words pronounced correctly
  Baseline - pre-injection | 100.0 (0.0)
  Baseline - post-injection | 87.0 (32.6)
  Week 2 - pre-injection: number analyzed (Participants) | 198
  Week 2 - pre-injection | 100.0 (0.0)
  Week 2 - post-injection: number analyzed (Participants) | 138
  Week 2 - post-injection | 91.7 (27.2)
  Week 4: number analyzed (Participants) | 195
  Week 4 | 100.0 (0.0)
  Week 8: number analyzed (Participants) | 197
  Week 8 | 100.0 (0.0)
  Week 12: number analyzed (Participants) | 179
  Week 12 | 100.0 (0.0)
  Week 16: number analyzed (Participants) | 180
  Week 16 | 100.0 (0.0)
  Week 24: number analyzed (Participants) | 182
  Week 24 | 100.0 (0.0)
  Week 36: number analyzed (Participants) | 173
  Week 36 | 100.0 (0.0)
  Week 52: number analyzed (Participants) | 46
  Week 52 | 100.0 (0.0)

10. Secondary Outcome: Assessments of the Lip Function by the Treating Investigator (TI) for the Safety Evaluation of TEOSYAL RHA® Redensity.
Description: as for outcome 9
Time Frame: as for outcome 9
Population: The following results reports data from subjects who received only the initial treatment (and if applicable, touch-up treatment) in order to confounding recovery with the effect of the new injection cycle(s).
Measure: Mean (Standard Deviation); unit: Proportion of touchpoints with sensation
Arm/Group | SAFT Population
Number analyzed (Participants) | 200
Proportion of touchpoints with sensation
  Baseline - pre-injection | 99.8 (2.4)
  Baseline - post-injection | 80.3 (36.0)
  Week 2 - pre-injection: number analyzed (Participants) | 198
  Week 2 - pre-injection | 100.0 (0.0)
  Week 2 - post-injection: number analyzed (Participants) | 138
  Week 2 - post-injection | 86.4 (32.11)
  Week 4: number analyzed (Participants) | 195
  Week 4 | 99.9 (1.19)
  Week 8: number analyzed (Participants) | 197
  Week 8 | 100.0 (0.0)
  Week 12: number analyzed (Participants) | 179
  Week 12 | 99.9 (1.3)
  Week 16: number analyzed (Participants) | 180
  Week 16 | 100.0 (0.0)
  Week 24: number analyzed (Participants) | 182
  Week 24 | 100.0 (0.0)
  Week 36: number analyzed (Participants) | 173
  Week 36 | 100.0 (0.0)
  Week 52: number analyzed (Participants) | 46
  Week 52 | 100.0 (0.0)

11. Secondary Outcome: Assessments of the Lip Function by the Treating Investigator (TI) for the Safety Evaluation of TEOSYAL RHA® Redensity.
Description: This Lip functionality testing was conducted by the Treating Investigator (TI) at each follow-up visit and pre- and post-injection at each injection, which occurred at Baseline, Weeks 2, 4, 8, 12, 16, 24, 36, and 52 after the last treatment. Lip sensation
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Proportion of touchpoints with sensation
Arm/Group | SAFT Population
Number analyzed (Participants) | 200
Proportion of touchpoints with sensation
  Baseline - pre-injection | 99.9 (1.2)
  Baseline - post-injection | 81.9 (35.4)
  Week 2 - pre-injection: number analyzed (Participants) | 198
  Week 2 - pre-injection | 100.0 (0.0)
  Week 2 - post-injection: number analyzed (Participants) | 138
  Week 2 - post-injection | 86.7 (31.9)
  Week 4: number analyzed (Participants) | 195
  Week 4 | 99.9 (1.19)
  Week 8: number analyzed (Participants) | 197
  Week 8 | 100.0 (0.0)
  Week 12: number analyzed (Participants) | 179
  Week 12 | 99.9 (1.25)
  Week 16: number analyzed (Participants) | 180
  Week 16 | 100.0 (0.0)
  Week 24: number analyzed (Participants) | 182
  Week 24 | 100.0 (0.0)
  Week 36: number analyzed (Participants) | 173
  Week 36 | 100.0 (0.0)
  Week 52: number analyzed (Participants) | 46
  Week 52 | 100.0 (0.0)

12. Other Pre Specified Outcome: Change From Baseline in Perioral Rhytids Severity Rating Scale (PR-SRS) Score Rated by the Treating Investigator (TI) at Weeks 4 and 8 After Last Treatment.
Description: The PR-SRS is a validated 4-point static scale for assessing perioral rhytids severity. Possible scores range from 0 (Absent) to 3 (Severe).
  Change = (Week 4 - Baseline score) and (Week 8 - Baseline score).
  A PR-SRS change of 1-grade will be considered clinically significant. The No-Treatment control group after treatment was not pooled for this exploratory outcome measure.
Time Frame: Weeks 4 and 8 after last treatment
Population: The Intent-to-Treat Population was used for this analysis. For this outcome measure, missing data were imputed using a LOCF (Last Observation Carried Forward) method.
Measure: Count of Participants; unit: Participants
Arm/Group | TEOSYAL RHA Redensity | No Treatment
Number analyzed (Participants) | 150 | 51
Participants
  Week 4: Responder | 145 | 2
  Week 4: Not Responder | 5 | 49
  Week 4: Missing values | 0 | 0
  Week 8: Responder | 143 | 1
  Week 8: Not Responder | 7 | 50
  Week 8: Missing values | 0 | 0

13. Other Pre Specified Outcome: Number of Subjects Scored Either "Much Improved" or "Improved" on Global Aesthetic Improvement (GAI) Scale by the Treating Investigator (TI) at Weeks 4 and 8 After Last Treatment.
Description: The Global Aesthetic Improvement (GAI) is a subjective, balanced, 5-point dynamic scale assessing cosmetic improvement.
  Possible scores range from "much improved", "improved", "no change", "worse", to "much worse".
  The GAI will be assessed using the pre-injection baseline photograph. The No-Treatment control group after treatment was not pooled for this exploratory outcome measure.
Time Frame: Weeks 4 and 8 after last treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TEOSYAL RHA Redensity | No Treatment
Number analyzed (Participants) | 150 | 51
Participants
  Week 4: Improved | 145 | 0
  Week 4: No Improvement | 1 | 48
  Week 4: Missing values | 4 | 3
  Week 8: Improved | 145 | 2
  Week 8: No Improvement | 2 | 47
  Week 8: Missing values | 3 | 2

14. Other Pre Specified Outcome: Change From Baseline of the Modified Glogau Classification of Wrinkling Rated by the Blinded Live Evaluator (BLE) at Week 8 After Last Treatment.
Description: The Modified Glogau Classification Scale is a 4-point classification measuring wrinkle severity. Possible scores range from 1 (Mild) to 4 (Severe).
  A Glogau score change of 1-grade will be considered clinically significant. The No-Treatment control group after treatment was not pooled for this exploratory outcome measure.
  Change = (Week 8 - Baseline score).
Time Frame: Week 8 after last treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TEOSYAL RHA Redensity | No Treatment
Number analyzed (Participants) | 150 | 51
Participants
  > or = 1-grade improvement from Baseline | 93 | 2
  < 1-grade improvement from Baseline | 53 | 46
  Missing values | 4 | 3

15. Other Pre Specified Outcome: Change From Baseline of the Modified Glogau Classification of Wrinkling Rated by the Treating Investigator (TI) at Weeks 4 and 8 After Last Treatment.
Description: The Modified Glogau Classification Scale is a 4-point classification measuring wrinkle severity. Possible scores range from 1 (Mild) to 4 (Severe).
  A Glogau score change of 1-grade will be considered clinically significant. The No-Treatment control group after treatment was not pooled for this exploratory outcome measure.
  Change = (Week 4 - Baseline score) and (Week 8 - Baseline score)
Time Frame: Weeks 4 and 8 after last treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TEOSYAL RHA Redensity | No Treatment
Number analyzed (Participants) | 150 | 51
Participants
  Week 4: > or = 1-grade improvement from Baseline | 105 | 2
  Week 4: < 1-grade improvement from Baseline | 41 | 46
  Week 4: Missing values | 4 | 3
  Week 8: > or = 1-grade improvement from Baseline | 106 | 4
  Week 8: < 1-grade improvement from Baseline | 41 | 45
  Week 8: Missing values | 3 | 2

16. Other Pre Specified Outcome: Change From Baseline in Perioral Rhytids Severity Rating Scale (PR-SRS) Score Rated by the Blinded Live Evaluator (BLE) at Weeks 8, 12, 16, 24, 36 and 52 After Last Treatment.
Description: The PR-SRS is a validated 4-point static scale for assessing perioral rhytids severity. Possible scores range from 0 (Absent) to 3 (Severe).
  Change = (Week 8 - Baseline score), (Week 12 - Baseline score), (Week 16 - Baseline score), (Week 24 - Baseline score), (Week 36 - Baseline score), (Week 52 - Baseline score)
  A PR-SRS change of 1-grade will be considered clinically significant. The No-Treatment control group after treatment was pooled for this exploratory outcome measure.
Time Frame: Weeks 8, 12, 16, 24, 36 and 52 after last treatment
Population: Of the randomized subjects (n=202), 2 subjects randomized to No-Treatment control did not receive treatment after the primary endpoint evaluation (Week 8 after randomization) and 1 subject randomized to No-Treatment control received treatment with study device, these 3 subjects are excluded from the pooled ITT population (n=199).
Measure: Count of Participants; unit: Participants
Groups:
- Intent-to-Treat Pooled Population: The ITT Pooled Population consisted of all the subjects randomized.
Arm/Group | Intent-to-Treat Pooled Population
Number analyzed (Participants) | 199
Participants
  Week 8: number analyzed (Participants) | 194
  Week 8: Responder | 156
  Week 8: Not Responder | 38
  Week 12: number analyzed (Participants) | 184
  Week 12: Responder | 156
  Week 12: Not Responder | 28
  Week 16: number analyzed (Participants) | 183
  Week 16: Responder | 147
  Week 16: Not Responder | 36
  Week 24: number analyzed (Participants) | 188
  Week 24: Responder | 137
  Week 24: Not Responder | 51
  Week 36: number analyzed (Participants) | 188
  Week 36: Responder | 131
  Week 36: Not Responder | 57
  Week 52: number analyzed (Participants) | 188
  Week 52: Responder | 125
  Week 52: Not Responder | 63

17. Other Pre Specified Outcome: Change From Baseline in Perioral Rhytids Severity Rating Scale (PR-SRS) Score Rated by the Treating Investigator (TI) at Weeks 4, 8, 12, 16, 24, 36 and 52 After Last Treatment.
Description: The PR-SRS is a validated 4-point static scale for assessing perioral rhytids severity. Possible scores range from 0 (Absent) to 3 (Severe).
  A PR-SRS change of 1-grade will be considered clinically significant. The No-Treatment control group after treatment was pooled for this exploratory outcome measure.
  Change = (Week 4 - Baseline score), (Week 8 - Baseline score), (Week 12 - Baseline score), (Week 16 - Baseline score), (Week 24 - Baseline score), (Week 36 - Baseline score), (Week 52 - Baseline score)
Time Frame: Weeks 4, 8, 12, 16, 24, 36 and 52 after last treatment
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Intent-to-Treat Pooled Population
Number analyzed (Participants) | 199
Participants
  Week 4: number analyzed (Participants) | 194
  Week 4: Responder | 187
  Week 4: Not Responder | 7
  Week 8: number analyzed (Participants) | 196
  Week 8: Responder | 186
  Week 8: Not Responder | 10
  Week 12: number analyzed (Participants) | 184
  Week 12: Responder | 175
  Week 12: Not Responder | 9
  Week 16: number analyzed (Participants) | 183
  Week 16: Responder | 171
  Week 16: Not Responder | 12
  Week 24: number analyzed (Participants) | 190
  Week 24: Responder | 173
  Week 24: Not Responder | 17
  Week 36: number analyzed (Participants) | 188
  Week 36: Responder | 161
  Week 36: Not Responder | 27
  Week 52: number analyzed (Participants) | 188
  Week 52: Responder | 149
  Week 52: Not Responder | 39

18. Other Pre Specified Outcome: Change From Baseline in Perioral Rhytids Severity Rating Scale (PR-SRS) Score Rated by Independent Photographic Reviewers (IPR) at Weeks 8, 12, 16, 24, 36 and 52 After Last Treatment.
Description: The PR-SRS is a validated 4-point static scale for assessing perioral rhytids severity. Possible scores range from 0 (Absent) to 3 (Severe).
  For a given subject to be considered a responder, at least 2 of the 3 readers must have confirmed a 1-point improvement for that subject The No-Treatment control group after treatment was pooled for this exploratory outcome measure.
  Change = (Week 8 - Baseline score), (Week 12 - Baseline score), (Week 16 - Baseline score), (Week 24 - Baseline score), (Week 36 - Baseline score), (Week 52 - Baseline score)
Time Frame: Weeks 8, 12, 16, 24, 36 and 52 after last treatment
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Intent-to-Treat Pooled Population
Number analyzed (Participants) | 199
Participants
  Week 8: number analyzed (Participants) | 196
  Week 8: Responder | 106
  Week 8: Not Responder | 90
  Week 12: number analyzed (Participants) | 183
  Week 12: Responder | 94
  Week 12: Not Responder | 89
  Week 16: number analyzed (Participants) | 177
  Week 16: Responder | 85
  Week 16: Not Responder | 92
  Week 24: number analyzed (Participants) | 188
  Week 24: Responder | 92
  Week 24: Not Responder | 96
  Week 36: number analyzed (Participants) | 186
  Week 36: Responder | 89
  Week 36: Not Responder | 97
  Week 52: number analyzed (Participants) | 188
  Week 52: Responder | 93
  Week 52: Not Responder | 95

19. Other Pre Specified Outcome: Change From Baseline of the Modified Glogau Classification of Wrinkling Rated by the Blinded Live Evaluator (BLE) at Week 8, 12, 16, 24, 36 and 52 After Last Treatment.
Description: The Modified Glogau Classification Scale is a 4-point classification measuring wrinkle severity. Possible scores range from 1 (Mild) to 4 (Severe).
  A Glogau score change of 1-grade will be considered clinically significant. The No-Treatment control group after treatment was pooled for this exploratory outcome measure.
  Change = (Week 8 - Baseline score), (Week 12 - Baseline score), (Week 16 - Baseline score), (Week 24 - Baseline score), (Week 36 - Baseline score), (Week 52 - Baseline score)
Time Frame: Weeks 8, 12, 16, 24, 36 and 52 after last treatment
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Intent-to-Treat Pooled Population
Number analyzed (Participants) | 199
Participants
  Week 8: number analyzed (Participants) | 194
  Week 8: > or = 1-grade improvement from Baseline | 117
  Week 8: < 1-grade improvement from Baseline | 77
  Week 12: number analyzed (Participants) | 184
  Week 12: > or = 1-grade improvement from Baseline | 116
  Week 12: < 1-grade improvement from Baseline | 68
  Week 16: number analyzed (Participants) | 183
  Week 16: > or = 1-grade improvement from Baseline | 112
  Week 16: < 1-grade improvement from Baseline | 71
  Week 24: number analyzed (Participants) | 188
  Week 24: > or = 1-grade improvement from Baseline | 99
  Week 24: < 1-grade improvement from Baseline | 89
  Week 36: number analyzed (Participants) | 188
  Week 36: > or = 1-grade improvement from Baseline | 93
  Week 36: < 1-grade improvement from Baseline | 95
  Week 52: number analyzed (Participants) | 188
  Week 52: > or = 1-grade improvement from Baseline | 89
  Week 52: < 1-grade improvement from Baseline | 99

20. Other Pre Specified Outcome: Change From Baseline of the Modified Glogau Classification of Wrinkling Rated by the Treating Investigator (TI) at Weeks 4, 8, 12, 16, 24, 36, and 52 After Last Treatment.
Description: The Modified Glogau Classification Scale is a 4-point classification measuring wrinkle severity. Possible scores range from 1 (Mild) to 4 (Severe).
  A Glogau score change of 1-grade will be considered clinically significant. The No-Treatment control group after treatment was pooled for this exploratory outcome measure.
  Change = (Week 4 - Baseline score), (Week 8 - Baseline score), (Week 12 - Baseline score), (Week 16 - Baseline score), (Week 24 - Baseline score), (Week 36 - Baseline score), (Week 52 - Baseline score)
Time Frame: Weeks 4, 8, 12, 16, 24, 36 and 52 after last treatment
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Intent-to-Treat Pooled Population
Number analyzed (Participants) | 199
Participants
  Week 4: number analyzed (Participants) | 194
  Week 4: > or = 1-grade improvement from Baseline | 135
  Week 4: < 1-grade improvement from Baseline | 59
  Week 8: number analyzed (Participants) | 196
  Week 8: > or = 1-grade improvement from Baseline | 134
  Week 8: < 1-grade improvement from Baseline | 62
  Week 12: number analyzed (Participants) | 184
  Week 12: > or = 1-grade improvement from Baseline | 129
  Week 12: < 1-grade improvement from Baseline | 55
  Week 16: number analyzed (Participants) | 183
  Week 16: > or = 1-grade improvement from Baseline | 117
  Week 16: < 1-grade improvement from Baseline | 66
  Week 24: number analyzed (Participants) | 190
  Week 24: > or = 1-grade improvement from Baseline | 115
  Week 24: < 1-grade improvement from Baseline | 75
  Week 36: number analyzed (Participants) | 188
  Week 36: > or = 1-grade improvement from Baseline | 106
  Week 36: < 1-grade improvement from Baseline | 82
  Week 52: number analyzed (Participants) | 188
  Week 52: > or = 1-grade improvement from Baseline | 85
  Week 52: < 1-grade improvement from Baseline | 103

21. Other Pre Specified Outcome: Subject's Perception of Treatment Effectiveness as Per the FACE-Q Scale (Perioral Rhytid Domain) Questionnaire at Week 4, 8, 12, 16, 24, 36, and 52 After Last Treatment.
Description: The FACE-Q measures the experience and outcomes of aesthetic facial procedures from the patient's perspective.
  The FACE-Q questionnaire is composed of 6 questions with a score linked to answers (1 being 'Not at all' and 4 being 'Extremely').
  To calculate the FACE-Q (Perioral Rhytids Domain) score, outcomes from all 6 questions were pooled, data were transformed so that higher scores reflected a superior (positive) outcome, and adapted to a scale of 100 units.
  The No-Treatment control group after treatment was pooled for this exploratory outcome measure.
Time Frame: Weeks 4, 8, 12, 16, 24, 36 and 52 after last treatment
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intent-to-Treat Pooled Population
Number analyzed (Participants) | 199
score on a scale
  Baseline Face-Q Score: number analyzed (Participants) | 198
  Baseline Face-Q Score | 22.8 (20.6)
  Week 4 Face-Q Score: number analyzed (Participants) | 194
  Week 4 Face-Q Score | 70.4 (22.8)
  Face-Q Change from Baseline to Week 4: number analyzed (Participants) | 193
  Face-Q Change from Baseline to Week 4 | 47.5 (26.9)
  Week 8 Face-Q Score: number analyzed (Participants) | 196
  Week 8 Face-Q Score | 69.3 (23.9)
  Face-Q Change from Baseline to Week 8: number analyzed (Participants) | 195
  Face-Q Change from Baseline to Week 8 | 46.5 (26.9)
  Week 12: number analyzed (Participants) | 184
  Week 12 | 68.3 (23.3)
  Face-Q Change from Baseline to Week 12: number analyzed (Participants) | 183
  Face-Q Change from Baseline to Week 12 | 45.4 (26.4)
  Week 16: number analyzed (Participants) | 182
  Week 16 | 66.8 (24.1)
  Face-Q Change from Baseline to Week 16: number analyzed (Participants) | 181
  Face-Q Change from Baseline to Week 16 | 43.4 (26.8)
  Week 24: number analyzed (Participants) | 190
  Week 24 | 62.0 (26.1)
  Face-Q Change from Baseline to Week 24: number analyzed (Participants) | 189
  Face-Q Change from Baseline to Week 24 | 38.9 (29.3)
  Week 36: number analyzed (Participants) | 188
  Week 36 | 62.1 (25.1)
  Face-Q Change from Baseline to Week 36: number analyzed (Participants) | 187
  Face-Q Change from Baseline to Week 36 | 38.8 (28.3)
  Week 52: number analyzed (Participants) | 188
  Week 52 | 59.0 (24.1)
  Face-Q Change from Baseline to Week 52: number analyzed (Participants) | 187
  Face-Q Change from Baseline to Week 52 | 36.2 (26.2)

22. Other Pre Specified Outcome: Number of Subjects Who Scored Themselves Either "Much Improved" or "Improved" on Global Aesthetic Improvement (GAI) Scale at Weeks 4, 8, 12, 16, 24, 36, 52 After Last Treatment.
Description: The Global Aesthetic Improvement (GAI) is a subjective, balanced, 5-point dynamic scale assessing cosmetic improvement.
  Possible scores range from "much improved", "improved", "no change", "worse", to "much worse".
  The GAI will be assessed using the baseline photograph. The No-Treatment control group after treatment was pooled for this exploratory outcome measure.
Time Frame: Weeks 4, 8, 12, 16, 24, 36 and 52 after last treatment
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Intent-to-Treat Pooled Population
Number analyzed (Participants) | 199
Participants
  Week 4: number analyzed (Participants) | 194
  Week 4: Improved | 191
  Week 4: No Improvement | 3
  Week 8: number analyzed (Participants) | 196
  Week 8: Improved | 186
  Week 8: No Improvement | 10
  Week 12: number analyzed (Participants) | 184
  Week 12: Improved | 165
  Week 12: No Improvement | 19
  Week 16: number analyzed (Participants) | 182
  Week 16: Improved | 162
  Week 16: No Improvement | 20
  Week 24: number analyzed (Participants) | 190
  Week 24: Improved | 158
  Week 24: No Improvement | 32
  Week 36: number analyzed (Participants) | 188
  Week 36: Improved | 152
  Week 36: No Improvement | 36
  Week 52: number analyzed (Participants) | 188
  Week 52: Improved | 156
  Week 52: No Improvement | 32

23. Other Pre Specified Outcome: Number of Subjects Scored Either "Much Improved" or "Improved" on Global Aesthetic Improvement (GAI) Scale by the Treating Investigator (TI) at Weeks 4, 8, 12, 16, 24, 36, 52 After Last Treatment.
Description: as for outcome 22
Time Frame: Weeks 4, 8, 12, 16, 24, 36 and 52 after last treatment.
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Intent-to-Treat Pooled Population
Number analyzed (Participants) | 199
Participants
  Week 4: number analyzed (Participants) | 194
  Week 4: Improved | 192
  Week 4: No Improvement | 2
  Week 8: number analyzed (Participants) | 196
  Week 8: Improved | 193
  Week 8: No Improvement | 3
  Week 12: number analyzed (Participants) | 184
  Week 12: Improved | 181
  Week 12: No Improvement | 3
  Week 16: number analyzed (Participants) | 183
  Week 16: Improved | 181
  Week 16: No Improvement | 2
  Week 24: number analyzed (Participants) | 190
  Week 24: Improved | 184
  Week 24: No Improvement | 6
  Week 36: number analyzed (Participants) | 188
  Week 36: Improved | 178
  Week 36: No Improvement | 10
  Week 52: number analyzed (Participants) | 188
  Week 52: Improved | 171
  Week 52: No Improvement | 17

24. Other Pre Specified Outcome: Number of Subjects Scored Either "Much Improved" or "Improved" on Global Aesthetic Improvement (GAI) Scale by the Blinded Live Evaluator (BLE) at Weeks 8, 12, 16, 24, 36, 52 After Last Treatment.
Description: as for outcome 22
Time Frame: Weeks 8, 12, 16, 24, 36 and 52 after last treatment
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Intent-to-Treat Pooled Population
Number analyzed (Participants) | 199
Participants
  Week 8: number analyzed (Participants) | 194
  Week 8: Improved | 179
  Week 8: No Improvement | 15
  Week 12: number analyzed (Participants) | 184
  Week 12: Improved | 166
  Week 12: No Improvement | 18
  Week 16: number analyzed (Participants) | 183
  Week 16: Improved | 160
  Week 16: No Improvement | 23
  Week 24: number analyzed (Participants) | 188
  Week 24: Improved | 158
  Week 24: No Improvement | 30
  Week 36: number analyzed (Participants) | 188
  Week 36: Improved | 156
  Week 36: No Improvement | 32
  Week 52: number analyzed (Participants) | 188
  Week 52: Improved | 152
  Week 52: No Improvement | 36

25. Other Pre Specified Outcome: Number of Subjects "Satisfied" or "Very Satisfied" With Study Treatment Using the Subject Satisfaction Scale at Weeks 4, 8, 12, 16, 24, 36, 52 After Last Treatment.
Description: The Subject Satisfaction Scale is a subjective, balanced, 5-point scale assessing subject satisfaction with study treatment. Possible scores range from with 1 (very satisfied) to 5 (very dissatisfied).
  The No-Treatment control group after treatment was pooled for this exploratory outcome measure.
Time Frame: Weeks 4, 8, 12, 16, 24, 36 and 52 after last treatment
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Intent-to-Treat Pooled Population
Number analyzed (Participants) | 199
Participants
  Week 4: number analyzed (Participants) | 194
  Week 4: Satisfied | 178
  Week 4: Not Satisfied | 16
  Week 8: number analyzed (Participants) | 196
  Week 8: Satisfied | 178
  Week 8: Not Satisfied | 18
  Week 12: number analyzed (Participants) | 183
  Week 12: Satisfied | 166
  Week 12: Not Satisfied | 17
  Week 16: number analyzed (Participants) | 182
  Week 16: Satisfied | 163
  Week 16: Not Satisfied | 19
  Week 24: number analyzed (Participants) | 190
  Week 24: Satisfied | 159
  Week 24: Not Satisfied | 31
  Week 36: number analyzed (Participants) | 188
  Week 36: Satisfied | 164
  Week 36: Not Satisfied | 24
  Week 52: number analyzed (Participants) | 188
  Week 52: Satisfied | 166
  Week 52: Not Satisfied | 22

26. Other Pre Specified Outcome: Number of Subjects With a Natural Look and Feel ≥7 of the Perioral Area, at Week 4, 8, 12, 16, 24, 36, and 52 After Last Treatment.
Description: The natural look and feel of the perioral area was assessed by subjects using an 11-point scale (ranging from 0 to 10).
  The No-Treatment control group after treatment was pooled for this exploratory outcome measure.
Time Frame: Weeks 8, 12, 16, 24, 36 and 52 after last treatment
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Intent-to-Treat Pooled Population
Number analyzed (Participants) | 199
Participants
  Baseline : Natural Look and Feel score > and = 7: number analyzed (Participants) | 198
  Baseline : Natural Look and Feel score > and = 7 | 91
  Week 4 : Natural Look and Feel score > and = 7: number analyzed (Participants) | 194
  Week 4 : Natural Look and Feel score > and = 7 | 171
  Week 8 : Natural Look and Feel score > and = 7: number analyzed (Participants) | 196
  Week 8 : Natural Look and Feel score > and = 7 | 174
  Week 12 : Natural Look and Feel score > and = 7: number analyzed (Participants) | 184
  Week 12 : Natural Look and Feel score > and = 7 | 164
  Week 16 : Natural Look and Feel score > and = 7: number analyzed (Participants) | 181
  Week 16 : Natural Look and Feel score > and = 7 | 158
  Week 24 : Natural Look and Feel score > and = 7: number analyzed (Participants) | 189
  Week 24 : Natural Look and Feel score > and = 7 | 158
  Week 36 : Natural Look and Feel score > and = 7: number analyzed (Participants) | 188
  Week 36 : Natural Look and Feel score > and = 7 | 160
  Week 52 : Natural Look and Feel score > and = 7: number analyzed (Participants) | 188
  Week 52 : Natural Look and Feel score > and = 7 | 164

27. Secondary Outcome: Assessments of the Lip Function by the Treating Investigator (TI) for the Safety Evaluation of TEOSYAL RHA® Redensity.
Description: as for outcome 9
Time Frame: as for outcome 9
Population: The following results reports data from subjects who received only the initial treatment (and if applicable, touch-up treatment), in order to confounding recovery with the effect of the new injection cycle(s).
Measure: Count of Participants; unit: Participants
Arm/Group | SAFT Population
Number analyzed (Participants) | 200
Participants
  Baseline - pre-injection: number analyzed (Participants) | 199
  Baseline - pre-injection: Able to use straw | 199
  Baseline - pre-injection: Not able to use straw | 0
  Baseline - post-injection: Able to use straw | 176
  Baseline - post-injection: Not able to use straw | 24
  Week 2 - pre-injection: number analyzed (Participants) | 198
  Week 2 - pre-injection: Able to use straw | 198
  Week 2 - pre-injection: Not able to use straw | 0
  Week 2 - post-injection: number analyzed (Participants) | 138
  Week 2 - post-injection: Able to use straw | 127
  Week 2 - post-injection: Not able to use straw | 11
  Week 4: number analyzed (Participants) | 195
  Week 4: Able to use straw | 195
  Week 4: Not able to use straw | 0
  Week 8: number analyzed (Participants) | 197
  Week 8: Able to use straw | 197
  Week 8: Not able to use straw | 0
  Week 12: number analyzed (Participants) | 179
  Week 12: Able to use straw | 179
  Week 12: Not able to use straw | 0
  Week 16: number analyzed (Participants) | 180
  Week 16: Able to use straw | 180
  Week 16: Not able to use straw | 0
  Week 24: number analyzed (Participants) | 182
  Week 24: Able to use straw | 182
  Week 24: Not able to use straw | 0
  Week 36: number analyzed (Participants) | 173
  Week 36: Able to use straw | 173
  Week 36: Not able to use straw | 0
  Week 52: number analyzed (Participants) | 46
  Week 52: Able to use straw | 46
  Week 52: Not able to use straw | 0

ADVERSE EVENTS:
Time Frame: - 52 to 58 (for patients receiving re-treatment) weeks for subjects randomized to TEOSYAL RHA® Redensity group. - 60 to 66 (for patients receiving re-treatment) weeks for subjects randomized to No-Treatment control group.
Groups:
- SAFT Population After Initial Treatment - V1/V1B to V9: The SAFT Population consisted of all subjects who were randomized and received at least one treatment with the study device during the course of the study (i.e. all subjects in the No-Treatment control group and all subjects in the TEOSYAL RHA® Redensity treatment group).
  Of the 202 randomized subjects, 2 subjects did not receive any treatment during the whole study, resulting in a SAFT population of n=200.
  For this pooled analysis, only AEs onset on or after initial study treatment are included : from V1/V1B to V9 (W52 or 56 weeks for patients receiving a re-treatment at W52). Therefore, for No-Treatment group, all AEs with onset date before initial treatment, i.e. V1b date, are excluded from this summary table.
- No Treatment - V1 to V4: No-Treatment group, before receiving initial treatment.
  For this pooled analysis, only AEs of subjects from the non-treatment group from V1(Baseline) to V4 (Week 8) are included.
- Treatment Group - V1 to V4: RHA Redensity group (Treatment group) from V1(Baseline) to V4 (Week 8) are included.
Arm/Group | SAFT Population After Initial Treatment - V1/V1B to V9 | No Treatment - V1 to V4 | Treatment Group - V1 to V4
All-Cause Mortality (participants affected / at risk) | 0/200 | 0/49 | 0/151
Serious Adverse Events (participants affected / at risk) | 7/200 | 0/49 | 1/151
Other Adverse Events (participants affected / at risk) | 120/200 | 7/49 | 74/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAFT Population After Initial Treatment - V1/V1B to V9 (N=200) | No Treatment - V1 to V4 (N=49) | Treatment Group - V1 to V4 (N=151)
Breast Cancer (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) — unrelated to the study device
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) — unrelated to the study device
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — unrelated to the study device
Pharyngeal Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — unrelated to the study device
Intraductal Proliferative Breast Lesion (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) — unrelated to the study device
Fallopian Tube Cancer (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) — unrelated to the study device
OTHER ADVERSE EVENTS (reported when occurring in more than 0.625% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAFT Population After Initial Treatment - V1/V1B to V9 (N=200) | No Treatment - V1 to V4 (N=49) | Treatment Group - V1 to V4 (N=151)
Blepharitis (Eye disorders) | 4 (4) | 3 (3) | 4 (5)
Vision Blurred (Eye disorders) | 3 (3) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Lip dry (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3)
Fatigue (General disorders) | 2 (2) | 1 (1) | 1 (1)
Injection site bruising (General disorders) | 23 (29) | 0 (0) | 14 (14)
Injection site discolouration (General disorders) | 14 (14) | 0 (0) | 5 (5)
Injection dryness (General disorders) | 2 (2) | 0 (0) | 2 (2)
Injection erythema (General disorders) | 10 (11) | 0 (0) | 4 (4)
Injection site hypoaesthesia (General disorders) | 4 (5) | 0 (0) | 2 (2)
Injection site induration (General disorders) | 22 (26) | 0 (0) | 13 (16)
Injection site mass (General disorders) | 34 (43) | 0 (0) | 25 (26)
Injection site movement impairment (General disorders) | 3 (3) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 14 (21) | 0 (0) | 10 (13)
Injection site pruritus (General disorders) | 6 (8) | 0 (0) | 5 (5)
Injection site scab (General disorders) | 2 (2) | 0 (0) | 2 (2)
Injection site swelling (General disorders) | 13 (16) | 0 (0) | 7 (7)
Influenza (Infections and infestations) | 5 (5) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 8 (8) | 0 (0) | 4 (4)
Oral Herpes (Infections and infestations) | 2 (3) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 29 (34) | 4 (4) | 20 (23)
Dizziness (Nervous system disorders) | 5 (6) | 1 (1) | 4 (4)
Needle track marks (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (1)
Skin wrinkling (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 2 (2)
Skin discolouration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1)
hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Needle track marks (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-10-27): https://cdn.clinicaltrials.gov/large-docs/19/NCT03092219/Prot_002.pdf
  • Statistical Analysis Plan (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT03092219/SAP_003.pdf